CLINICAL TRIAL: NCT01909089
Title: Determination of the Minimum Local Analgesic Dose of Spinal Chloroprocaine in Labour.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/334; 2013-001703-37 (EudraCT Number)
Record Dates: First submitted 2013-07-23; First posted 2013-07-26 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Pain Relief During Labour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chloroprocaine (Experimental): Up-down sequential allocation.
  Interventions: Drug: Spinal administration of chloroprocaine.

INTERVENTIONS:
Drug: Spinal administration of chloroprocaine. — In order to determine the minimum effective dose that is to be given spinally, an up-down sequential allocation will be used.
  Efficacy of the analgesia will be evaluated by a 100mm visual analogue pain score (VAPS). There are two possible outcomes here:
  * effective: the VAPS is 10mm or lower after the 15 minutes of monitoring. An effective result will decrease the test dose of chloroprocaine with 2mg for the next patient in this study.
  * Ineffective: the VAPS is more than 10mm after 15 minutes of monitoring. An ineffective result will increase the test dose of chloroprocaine with 2mg for the next patient in this study. Patients who indicate an ineffective result will receive a rescue treatment by the administration of 12ml levobupivacaine epidurally.

SUMMARY:
Combined spinal-epidural (CSE) analgesia has become a widely accepted approach to provide analgesia for labour pain. Despite the increasingly widespread use of this technique, an optimal intrathecal drug regimen has not been established yet.

Several investigations using local anesthetics such as Bupivacaine, Levobupivacaine and Ropivacaine in CSE during labour have been published. But despite the reintroduction of Chloroprocaine recently there haven't been any investigations about spinal chloroprocaine. Chloroprocaine is already a long-know drug with a beneficial pharmacodynamic/kinetic profile. It is known for a very quick onset of action (2 - 3 minutes), high efficacy, rapid metabolism by plasma cholinesterases and short half-life both in mother and fetus.

Because of this beneficial profile, Chloroprocaine is widely used intrathecally for surgical anesthesia. Several investigations demonstrate that for surgical anesthesia doses Chloroprocaine ranging from 30 - 60 mg are used and that they have an effective surgical duration of 40 - 90 minutes.

Despite these "standards" for surgical anesthesia, little is known about spinal Chloroprocaine dose regimens. Therefore the primary goal of this study is to determine the minimum adequate dose of Chloroprocaine that is to be given spinally to a woman in labour using a CSE procedure. We will use the up-down sequential allocation to identify the median effective dose (ED50) or concentration (EC50).

The Effective dose in 95% of the population (ED95) can be estimated also from an up-down sequential allocation and will become an important valuable approximation of the clinical dose.

ELIGIBILITY:
Inclusion criteria :

* Pregnant women in labour with a gestational period of 36 to 41 weeks
* ASA I or II
* Primi- and multiparae
* Spontaneous or induced labor

Exclusion criteria :

Pregnant women in labour who received opiates or analgetics during the 6 hour period prior to CSE

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2015-08-21 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Intensity of sensory blockade during the next 15 minutes after the application of the CSE. | During the next 15 minutes after the application of the CSE.
  The sensory blockade is determined by the difference in temperature sensation over the different dermatomes aided by ethylchloride spray.
Intensity of the motor blockade during the next 15 minutes after the application of the CSE. | During the next 15 minutes after the application of the CSE.
  The motor blockade is determined by the adjusted Bromage scale:
  1. = complete motor block with the impossibility to move the legs
  2. = only the possibility to move the feet
  3. = possibility to move the knees
  4. = weak flexion of the hips
  5. = a complete flexion of the hips and the knees
  Prior to the application of the CSE the patients are asked to perform the motor tests to exclude neurological disorders.
The analgesic effect on the labor pain during the next 15 minutes after the application of the CSE. | During the next 15 minutes after the application of the CSE.
  Efficacy of the analgesia will be evaluated by a 100mm visual analogue pain score (VAPS). There are two possible outcomes here:
  * effective: the VAPS is 10mm or lower after the 15 minutes of monitoring. An effective result will decrease the test dose of chloroprocaine with 2mg for the next patient in this study.
  * Ineffective: the VAPS is more than 10mm after 15 minutes of monitoring. An ineffective result will increase the test dose of chloroprocaine with 2mg for the next patient in this study. Patients who indicate an ineffective result will receive a rescue treatment by the administration of 12ml levobupivacaine epidurally.

SECONDARY OUTCOMES:
Maternal heart rate during application of the CSE and the hour there after. | During application of the CSE and the hour there after.
Maternal blood pressure during application of the CSE and the hour there after. | During application of the CSE and the hour there after.
Maternal oxygen saturation during application of the CSE and the hour there after. | During application of the CSE and the hour there after.
Fetal heart rate during application of the CSE and the hour there after. | During application of the CSE and the hour there after.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Coppens, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be